CLINICAL TRIAL: NCT00098358
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Clinical Proof of Concept Study of Zileuton IR in Patients With Moderate to Severe Facial Acne Vulgaris
Brief Title: Study of Oral Zileuton in the Treatment of Moderate to Severe Facial Acne Vulgaris
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Critical Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTI-02-C04-201
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2007-02-07 (Estimated); Status verified 2007-02

CONDITIONS: Acne Vulgaris
Keywords: Leukotrienes; inflammation
MeSH Terms: conditions — Acne Vulgaris; Inflammation | interventions — zileuton

INTERVENTIONS:
Drug: Zileuton

SUMMARY:
Tissue inflammation is a major component of the acne disease process. Leukotriene B4 (LTB4) is thought to be a major player in the development of tissue inflammation. Synthesis of LTB4 is controlled by the enzyme 5-lipoxygenase. Zileuton blocks the activity of 5-lipoxygenase. This study will test the safety and efficacy of zileuton in the treatment of facial acne.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe facial acne vulgaris
* 20 to 60 facial inflammatory lesions
* 10 to 200 facial non-inflammatory lesions
* No more than 3 facial nodular cystic lesions

Exclusion Criteria:

* Uncontrolled systemic disease
* Use of systemic or topical acne therapy within 14 days of study
* Use of systemic retinoids within past 2 years
* Skin diseases that interfere with acne counts
* Active liver disease
* Screening elevations in liver function tests
* Positive serology for hepatitis B or C
* Use of theophylline, warfarin, or propranolol within 7 days of study
* Use of Singulair or Accolate within 14 days of study
* Female patients who are pregnant or nursing

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2004-11; Study Completion 2005-05

PRIMARY OUTCOMES:
Change in number of inflammatory lesions

SECONDARY OUTCOMES:
Physician's global assessment scale
Change in number of non-inflammatory lesions
Change in total numbers of lesions
Change in sebum production

CONTACTS AND LOCATIONS:
Overall Officials: Walter Newman, Ph.D., Study Director — Critical Therapeutics
Locations (12):
- United States (12):
  - Therapeutics Clinical Research, San Diego, California
  - MedaPhase, Inc., Newnan, Georgia
  - Dermatology Specialists, PSC, Louisville, Kentucky
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Dermatology Associates of Rochester, Rochester, New York
  - Milton S. Hersey Medical Center, Hersey, Pennsylvania
  - Rivergate Dermatology, Goodlettsville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - J&S Studies, Inc., Bryan, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

REFERENCES:
- [Background] Zouboulis CC, Nestoris S, Adler YD, Orth M, Orfanos CE, Picardo M, Camera E, Cunliffe WJ. A new concept for acne therapy: a pilot study with zileuton, an oral 5-lipoxygenase inhibitor. Arch Dermatol. 2003 May;139(5):668-70. doi: 10.1001/archderm.139.5.668. No abstract available. PMID 12756111